CLINICAL TRIAL: NCT00613262
Title: A Prospective, Single Blinded Study for Predicting Colon Polyp Histology With Narrow Band Imaging
Acronym: NBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Midwest Biomedical Research Foundation (Other)
Responsible Party: Principal Investigator, Amit Rastogi, Principal Investagator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: AR0002; 00371
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2009-02

CONDITIONS: Colonoscopy; Adenomatous Polyp; Neoplastic
Keywords: Narrow Band Imaging
MeSH Terms: conditions — Adenomatous Polyps | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Narrow Band Imaging — Narrow Band Imaging Colonoscope offers an alternative lightsource to view colon polyps in real time

SUMMARY:
The investigators hypothesize that NBI will have a high accuracy in predicting polyp histology real time during a colonoscopy by visualization of the surface mucosal and vascular patterns. Aim#1: To determine the sensitivity, specificity and accuracy of NBI and standard white light colonoscopy for predicting polyp histology by evaluating the surface mucosal and vascular patterns during colonoscopy. Aim#2: To determine the inter-observer agreement between investigators for the recognition of various polyp patterns.

ELIGIBILITY:
Inclusion Criteria:

* referral for screening or surveillance colonoscopy
* the ability to provide informed consent

Exclusion Criteria:

* prior surgical resection of any portion of colon
* prior history of colon cancer
* history of inflammatory bowel disease
* use of anti-platelet agents or anticoagulants that precludes removal of polyps during the procedure
* poor general condition or any other reason to avoid prolonged procedure time
* history of polyposis syndrome or Hereditary Non-polyposis colon cancer
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The mucosal and vascular patterns and their correlation with polyp histology will be used as the primary outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amit Rastogi, MD, Principal Investigator — Kansas City VA Medical Center
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States